CLINICAL TRIAL: NCT03862534
Title: Coronally Advanced Flap (CAF) and Composite Restoration of the Enamel With or Without Connective Tissue Graft (CTG) for the Treatment of Single Maxillary Gingival Recession With Non-carious Cervical Lesion (NCCL). A Randomized Controlled Clinical Trial
Brief Title: CAF With or Without CTG for the Treatment of Single Maxillary Gingival Recession With NCCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Dr. Francesco Cairo, Head, Research Unit in Periodontology and Periodontal Medicine, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT restored CEJ
Record Dates: First submitted 2019-02-27; First posted 2019-03-05 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Gingival Recession
Keywords: Gingival recession; Non-carious cervical lesion; Connective tissue graft
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAF (Experimental): After the restoration of the enamel patients were treated with a CAF
  Interventions: Procedure: CAF
- CAF + CTG (Experimental): After the restoration of the enamel patients were treated with a CAF + CTG
  Interventions: Procedure: CAF + CTG

INTERVENTIONS:
Procedure: CAF — After the cementum enamel junction (CEJ) was restorated, a split thickness flap was raised, coronally advanced and sutured to cover the recession
  Arms: CAF
Procedure: CAF + CTG — After the cementum enamel junction (CEJ) was restorated, a split thickness flap was raised. Then a connective tissue graft was harvested from the palate and sutured over the exposed root. Finally the flap was coronally advanced and sutured to cover the recession
  Arms: CAF + CTG

SUMMARY:
This studies evaluate the efficacy of the coronally advanced flap (CAF) with or without connective tissue graft (CTG) for the treatment of single maxillary recession associated to non carious cervical lesion (NCCL).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* No systemic diseases or pregnancy.
* Self-reported smoking ≤ 10 cigarettes/day.
* Full-mouth plaque score (FMPS) and full-mouth bleeding score (FMBS) ≤ 10% (measured at four sites per tooth).
* Presence of single RT1 buccal gingival recessions ≥ 2 mm of depth located in the anterior area of the upper jaw (central and lateral incisors, canine, first and second pre-molars, first molar) and associated with aesthetic complains and or dental sensitivity.
* Presence of NCCL associated with recession
* No history of mucogingival or periodontal surgery at experimental sites.

Exclusion Criteria:

* Prosthetic crown at experimental teeth.
* Gingival recessions presenting minimal amount (< 1mm) of apico-coronal keratinized tissue (KT) extension apical to recession area.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Recession Reduction | At 12 months
  Difference between gingival recession at 12 months and baseline, measured with a periodontal probe.
Complete Root Coverage (CRC) | At 12 months
  Absence or presence of gingival recession at 12 months follow-up.

SECONDARY OUTCOMES:
Root coverage Esthetic Score (RES) | At 12 months
  Overall esthetic score from 0 to 10 evaluated by the blinded examiner. Higher values represent a better outcome. (Pini-Prato et al. 2011)
Gingival Thickness (GT) | Baseline - 12 months
  Gingival thickness in mm, measured with an endodontic file and a digital caliper.
Keratinized Tissue (KT) | Baseline - 6 and 12 months
  Width of the keratinized gingiva measured in mm from the gingival margin to the muco-gingival-junction using a periodontal probe
KTgain | At 12 months
  Gain of Keratinized Tissue measured as the difference between KT at 12 months and KT baseline
Gingival Recesión (REC) | Baseline - 6 and 12 months
  The distance between the reconstructed cementum enamel junction and the gingival margin measured in mm with a periodontal probe
Root sensitivity | Baseline - 6 and 12 months
  Toot sensitivity reported by the patient present or absent
SensVAS | Baseline - 6 and 12 months
  Toot sensitivity reported by the patient on a 0 to 10 Visual Analogue Scale. Higher values represent worse outcome.
SurTime | At surgery
  Surgical Time in minutes from the end of anesthesia to the sutures
Anti-infammTab | 1 week post-surgery
  Number of tablets of anti-inflammatory drug taken in the first week post-operatively by the patients.
DiscVAS | 1 week post-surgery
  Post Operative Discomfort reported by the patients on a 0 to 10 Visual Analogue Scale. Higher values represent worse outcome.
AesthVAS | At 12 months
  Aesthetic overall satisfaction reported by the patients on a 0 to 10 Visual Analogue Scale. Higher values represent better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cairo, DDS, Principal Investigator — University of Florence

REFERENCES:
- [Background] Cairo F. Periodontal plastic surgery of gingival recessions at single and multiple teeth. Periodontol 2000. 2017 Oct;75(1):296-316. doi: 10.1111/prd.12186. PMID 28758301
- [Background] Cairo F, Pagliaro U, Buti J, Baccini M, Graziani F, Tonelli P, Pagavino G, Tonetti MS. Root coverage procedures improve patient aesthetics. A systematic review and Bayesian network meta-analysis. J Clin Periodontol. 2016 Nov;43(11):965-975. doi: 10.1111/jcpe.12603. Epub 2016 Sep 16. PMID 27454460
- [Background] Cairo F, Pini-Prato GP. A technique to identify and reconstruct the cementoenamel junction level using combined periodontal and restorative treatment of gingival recession. A prospective clinical study. Int J Periodontics Restorative Dent. 2010 Dec;30(6):573-81. PMID 20967303
- [Background] Hwang D, Wang HL. Flap thickness as a predictor of root coverage: a systematic review. J Periodontol. 2006 Oct;77(10):1625-34. doi: 10.1902/jop.2006.060107. PMID 17032103
- [Background] Cortellini P, Tonetti M, Baldi C, Francetti L, Rasperini G, Rotundo R, Nieri M, Franceschi D, Labriola A, Prato GP. Does placement of a connective tissue graft improve the outcomes of coronally advanced flap for coverage of single gingival recessions in upper anterior teeth? A multi-centre, randomized, double-blind, clinical trial. J Clin Periodontol. 2009 Jan;36(1):68-79. doi: 10.1111/j.1600-051X.2008.01346.x. Epub 2008 Nov 20. PMID 19046326
- [Background] Santamaria MP, da Silva Feitosa D, Nociti FH Jr, Casati MZ, Sallum AW, Sallum EA. Cervical restoration and the amount of soft tissue coverage achieved by coronally advanced flap: a 2-year follow-up randomized-controlled clinical trial. J Clin Periodontol. 2009 May;36(5):434-41. doi: 10.1111/j.1600-051X.2009.01389.x. PMID 19419445
- [Background] Zucchelli G, Gori G, Mele M, Stefanini M, Mazzotti C, Marzadori M, Montebugnoli L, De Sanctis M. Non-carious cervical lesions associated with gingival recessions: a decision-making process. J Periodontol. 2011 Dec;82(12):1713-24. doi: 10.1902/jop.2011.110080. Epub 2011 May 4. PMID 21542735